CLINICAL TRIAL: NCT05922059
Title: Effects of Autonomic Nervous System Modulation on Heart Rate Variability and Musculoskeletal Manifestations in Patients With Chronic Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Hani Alkhawajah, Principal Investigator - Senior Physiotherapist, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-PGS-2023-03-096
Record Dates: First submitted 2023-06-08; First posted 2023-06-28 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Autonomic Nervous System Modulation
Keywords: Vagus nerve stimulation; Neck pain; Heart rate variability; Heart rhythm coherence feedback
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: Group A (transcutaneous vagus nerve stimulation + standard-care physiotherapy), Group B (HRV-BF + standard-care physiotherapy), or Group C (standard-care physiotherapy alone).
Who Masked: Participant, Outcomes Assessor
Masking Description: A receptionist will inform the treating therapist about the patient's allocation later after the baseline measurements are performed.
  An independent, a physiotherapist (assessor) from the Department of Physiotherapy (with > 10 years of clinical experience in physiotherapy) who is blinded to the allocation (treatment group) of the patients will collect the demographic data and baseline outcome measurements. Then, the assessor will leave the room to remain blind to conditions. At the same time, the treating physiotherapist, the main researcher, (with > 10 years of clinical experience in musculoskeletal physiotherapy) will apply the treatment protocol according to the patient's allocated group. The treating therapist will be blind to the outcome measurements until the patients end their role in the study. Patients will be asked not to discuss their treatment experience with the assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vagus nerve stimulation (Experimental): Transcutaneous vagus nerve stimulation in addition to standard-care physiotherapy
  Interventions: Device: Transcutaneous vagus nerve stimulation
- Heart rate variability biofeedback (Experimental): Heart rate variability biofeedback in addition to standard-care physiotherapy
  Interventions: Device: Heart rate variability biofeedback
- standard-care physiotherapy alone (Active Comparator): standard-care physiotherapy
  Interventions: Other: Standard-care physiotherapy

INTERVENTIONS:
Device: Transcutaneous vagus nerve stimulation — Auricular transcutaneous vagus nerve stimulation will be used in the left cavity of the external ear with a stimulation frequency of 20-30 Hz for half hour. Monophasic rectangular waveforms will be used, and the intensity will be adjusted below the patient's pain threshold.
  Arms: Vagus nerve stimulation
Device: Heart rate variability biofeedback — The patient will receive visual HRV feedback during resonance frequency breathing. Finally, the patient will be instructed to maximize their peak-to-peak HRV and attain the phase between respiration and HRV changes as closely as possible
  Arms: Heart rate variability biofeedback
Other: Standard-care physiotherapy — consists of cervical mobilization on the painful segment, isometric exercise for neck flexors, and a combination of strengthening and stretching exercises from sitting position; cervical extensors strengthening exercise using red color Thera-band and stretching exercises upper trapezius of the painful side.
  Arms: standard-care physiotherapy alone

SUMMARY:
Background: Chronic neck pain is a widespread musculoskeletal disorder. Studies investigating the effect of autonomic nervous system (ANS) modulation in chronic neck pain are scarce. This study aims to examine the effects of ANS modulation on heart rate variability, pain, and function in patients with chronic neck pain. Methods: The intended study is a double-blind, randomized controlled trial in a parallel three arms fashion. Hundred and two patients with chronic neck pain will be recruited from King Fahd Hospital of the University in Alkhobar, Saudi Arabia. The patients will be randomly allocated equally into one of three groups. Group A (n = 34) will receive transcutaneous vagus nerve stimulation (tVNS) and standard-care physiotherapy (SC-PT). Group B (n = 34) will receive heart rate variability biofeedback (HRV-BF) and SC-PT. Group C (n = 34) will receive SC-PT alone. Each group will receive the intervention three times per week for six weeks. The primary outcome measures are HRV to assess ANS and the visual analog scale for pain intensity. The secondary outcome measures are pressure pain threshold and neck disability index. All these measures will be assessed on three occasions; at baseline, after three weeks, and after six weeks from baseline. For the statistical analysis, normality of the data will be performed prior to the analyses and suitable statistical tests will be applied to examine the effect of the interventions between the groups. The significance level sets at P < 0.05.

DETAILED DESCRIPTION:
Sample size calculation was performed using statistical software (G*Power 3.1). The effect size (ES) of HRV was obtained from a previous study (Hallman et al., 2011). The following combination was used to calculate the sample size: analysis of variance (ANOVA), repeated measures, within-between interaction, ES of 0.15, an alpha level of 0.05, power (1-β) of 80%, correlation among repeated measure of 0.5, with three groups and three measurements (time points) and non-sphericity correction (Є) of 1. The estimated desired sample size was 93 patients. Three patients per group will be needed considering a 10% attrition rate. Thus, the total required sample size is 102 patients, 34 patients in each group.

The study will be conducted in the Department of Physiotherapy at KFHU Saudi Arabia. Patients with chronic neck pain who will attend KFHU and fit the inclusion criteria will be recruited consecutively and randomly allocated into Group A (transcutaneous vagus nerve stimulation + standard-care physiotherapy), Group B (HRV-BF + standard-care physiotherapy), or Group C (standard-care physiotherapy alone). The randomization sequence will be computer-generated using the GraphPad website (http://www.graphpad.com/). Hundred and two patients will be uniquely randomized equally into three different groups; each number and its allocated group will be written on a piece of paper and concealed in an opaque envelope. A receptionist will inform the treating therapist about the patient's allocation later after the baseline measurements are performed.

An independent, a physiotherapist (assessor) from the Department of Physiotherapy (with > 10 years of clinical experience in physiotherapy) who is blinded to the allocation (treatment group) of the patients will collect the demographic data and baseline outcome measurements. Then, the assessor will leave the room to remain blind to conditions. At the same time, the treating physiotherapist, the main researcher, (with > 10 years of clinical experience in musculoskeletal physiotherapy) will apply the treatment protocol according to the patient's allocated group. The treating therapist will be blind to the outcome measurements until the patients end their role in the study. Patients will be asked not to discuss their treatment experience with the assessor. The assessor will perform the outcome measurements three weeks and six weeks after intervention.

ELIGIBILITY:
Inclusion Criteria:

* adult aged ≥ 18 years old
* have had neck pain for three months or more
* reported peak neck pain of more than three on visual analogue scale (VAS) over the previous 24 hours

Exclusion Criteria:

* have had neck surgery
* intra-articular corticosteroid injection within six months
* current or past (within four weeks) oral corticosteroid use
* neurological conditions
* altered sensation to pressure
* pregnancy
* exhibited cognitive difficulties
* arm numbness or tingling
* cardiac pacemaker or other implantable stimulators
* cardiac arrhythmia
* history of myocardial infarction
* local auricular diseases
* symptomatic orthostatic hypotension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2023-07-18 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart-rate variability (HRV) | Baseline
  the changes in the inter-beat intervals (IBIs) that will be used to quantify the amount of HRV observed during monitoring periods (<1 min to >24 h). In this study, the monitoring period will be five minutes
Heart-rate variability (HRV) | Change from baseline HRV after 3 weeks
  the changes in the inter-beat intervals (IBIs) that will be used to quantify the amount of HRV observed during monitoring periods (<1 min to >24 h). In this study, the monitoring period will be five minutes
Heart-rate variability (HRV) | Change from baseline HRV after 6 weeks
  the changes in the inter-beat intervals (IBIs) that will be used to quantify the amount of HRV observed during monitoring periods (<1 min to >24 h). In this study, the monitoring period will be five minutes
Visual analog scale (VAS) | Baseline
  Current pain intensity will be measured using a 10-cm VAS with endpoints marked 'no pain' at 0 and 'worst pain imaginable at 10.
Visual analog scale (VAS) | Change from baseline VAS after 3 weeks
  Current pain intensity will be measured using a 10-cm VAS with endpoints marked 'no pain' at 0 and 'worst pain imaginable at 10.
Visual analog scale (VAS) | Change from baseline VAS after 6 weeks
  Current pain intensity will be measured using a 10-cm VAS with endpoints marked 'no pain' at 0 and 'worst pain imaginable at 10.

SECONDARY OUTCOMES:
Pressure pain threshold (PPT) | Baseline
  A digital pressure algometer (Somedic AB, Farsta, Sweden) with a surface probe of 1 cm2 and a rate of 40 kPa/s will be used to quantify the pain intensity. The measurement will be taken on the painful area. Participants will be instructed to activate a button when the sensation of pressure becomes painful, and the resultant value will be recorded. Three measurements will be performed. The average value will be recorded for analysis.
Pressure pain threshold (PPT) | Change from baseline PPT after 3 weeks
  A digital pressure algometer (Somedic AB, Farsta, Sweden) with a surface probe of 1 cm2 and a rate of 40 kPa/s will be used to quantify the pain intensity. The measurement will be taken on the painful area. Participants will be instructed to activate a button when the sensation of pressure becomes painful, and the resultant value will be recorded. Three measurements will be performed. The average value will be recorded for analysis.
Pressure pain threshold (PPT) | Change from baseline PPT after 6 weeks
  A digital pressure algometer (Somedic AB, Farsta, Sweden) with a surface probe of 1 cm2 and a rate of 40 kPa/s will be used to quantify the pain intensity. The measurement will be taken on the painful area. Participants will be instructed to activate a button when the sensation of pressure becomes painful, and the resultant value will be recorded. Three measurements will be performed. The average value will be recorded for analysis.
Neck Disability Index (NDI) | Baseline
  The NDI is a self-assessment questionnaire for the specific functional status of individuals with neck pain. It consists of ten sections: pain, personal care, weight gain, reading, headache, concentration, work, driving, sleeping, and leisure. Each section is scaled from 0 to 5, where 0 represents "painless" and 5 represents "the worst pain imaginable." The points obtained are added to a total score.
Neck Disability Index (NDI) | Change from baseline NDI after 3 weeks
  The NDI is a self-assessment questionnaire for the specific functional status of individuals with neck pain. It consists of ten sections: pain, personal care, weight gain, reading, headache, concentration, work, driving, sleeping, and leisure. Each section is scaled from 0 to 5, where 0 represents "painless" and 5 represents "the worst pain imaginable." The points obtained are added to a total score.
Neck Disability Index (NDI) | Change from baseline NDI after 6 weeks
  The NDI is a self-assessment questionnaire for the specific functional status of individuals with neck pain. It consists of ten sections: pain, personal care, weight gain, reading, headache, concentration, work, driving, sleeping, and leisure. Each section is scaled from 0 to 5, where 0 represents "painless" and 5 represents "the worst pain imaginable." The points obtained are added to a total score.

IPD SHARING:
Plan to Share IPD: Yes
The work will be published in peer review journal
Supporting Information: Study Protocol, SAP
Time Frame: When data collection finalized. A manuscript will be written for publication. The estimated time is 1 year. After publication in peer review journal, the data will remain in the journal in accordance to journal policy